CLINICAL TRIAL: NCT07129356
Title: Feasibility a Combining Rehabilitation Program at Field Exercises and Tele-exercises to Enhance Daily Life Activities to Rural Women in Iraq
Brief Title: Field and Home Exercise Program for Improving Function in Iraqi Rural Women
Acronym: CRP-Rural
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mosul (Other)
Responsible Party: Principal Investigator, Munib Abdullah Fathi, Assistant Professor Doctorate, University of Mosul
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: College of Physical Education; The corresponding Author (Other: University of Mosul)
Record Dates: First submitted 2025-07-23; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Rural Health; Physical Therapy; Rehabilitation
Keywords: Muscle imbalance; Chronic musculoskeletal pain; Back pain
MeSH Terms: conditions — Chronic Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: Design: Quasi-Experimental, One-Group Pretest-Posttest Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Rehabilitation Program (CRP) - Single Group (Experimental): This arm received a 12-week Combined Rehabilitation Program (CRP), consisting of both in-person field exercises and remote tele-exercises. The intervention included therapeutic exercises and culturally relevant physical games tailored to improve musculoskeletal function and reduce pain. Exercises were focused on mobility, strength, and flexibility, targeting areas of muscle weakness identified during baseline assessment.
  Interventions: Behavioral: Combined Exercise

INTERVENTIONS:
Behavioral: Combined Exercise — Participants engaged in a hybrid exercise program that included:
  In-field sessions held twice weekly at a local sports facility (45-60 minutes per session, including rest).
  Remote sessions delivered via pre-recorded videos through WhatsApp, with ongoing monitoring and feedback.
  Exercises included walking, jogging, full-body stretching, and strength training targeting the trunk, limbs, and weak muscle groups (shoulders, back, knees).
  The program aimed to reduce joint and muscle pain, improve strength and flexibility, and support daily functional activities.
  Pre- and post-intervention assessments included muscle strength (via hand dynamometer), flexibility tests, BMI, and self-reported pain using the NRS-11 scale.

SUMMARY:
This study evaluates a 12-week Combined Rehabilitation Program (CRP) designed to reduce musculoskeletal pain and improve physical function among rural women in northern Iraq. The program integrates home-based therapeutic exercises with simple, culturally appropriate games. Sixty-six women from the Hamdaniya district, all with nearly two decades of experience in agricultural labor and chronic musculoskeletal pain in the back, neck, and limbs, participated voluntarily.

The intervention includes two supervised group sessions per week at a local sports field and remote home-based sessions guided via pre-recorded videos shared through WhatsApp. Each session lasts 45 to 60 minutes and incorporates rest periods. The program is designed to strengthen weakened muscles, improve daily function, and promote social engagement among participants.

Rural women engaged in long-term agricultural labor are at increased risk of chronic musculoskeletal pain, particularly in the back, neck, and limbs.

What is already known on this subject:

* Rural women engaged in long-term agricultural labor are at increased risk of chronic musculoskeletal pain, particularly in the back, neck, and limbs.
* Home-based therapeutic exercises are widely used to manage pain and improve physical function.
* Community-based rehabilitation programs can support better health outcomes in underserved populations.

What this study adds:

* Introduces a culturally adapted Combined Rehabilitation Program (CRP) that blends home-based exercises with traditional games in a rural Iraqi context.
* Explores the feasibility of delivering rehabilitation through low-cost mobile technology in resource-limited environments.
* Provides a community-based model for accessible, flexible rehabilitation tailored to the needs of rural women.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of a Combined Rehabilitation Program (CRP) designed to reduce musculoskeletal pain and enhance physical function among rural women in northern Iraq. The CRP integrates home-based therapeutic exercises with culturally relevant physical games and is tailored to the specific needs and social context of the participants.

The study includes 66 women, aged around 46 years, with 18-23 years of experience in agricultural work. All participants reported ongoing muscle and joint pain in the upper and lower limbs, back, and neck, which affects their ability to carry out daily activities. Due to family and work constraints, a flexible intervention was developed that combines in-person and remote elements to ensure accessibility and adherence.

The 12-week program consists of two supervised group sessions per week held at a local field, along with home-based sessions delivered through pre-recorded videos shared via mobile applications. Each session lasts 45-60 minutes and includes walking, stretching, strengthening exercises, and simple games targeting muscle groups commonly affected by physical labor. Rest periods are integrated into each session to promote safety and participation.

Participants are assessed before and after the intervention for muscle strength, flexibility, body composition, and pain levels using standardized tools. The study design emphasizes a community-based and technology-supported approach to rehabilitation, addressing the unique challenges faced by women in rural areas with limited access to conventional services.

ELIGIBILITY:
Inclusion Criteria:

* Women have experienced Musculoskeletal pain in one or more one of fourth areas of study variables which are : the upper and lower extremities, neck, and lower back.

Exclusion Criteria:

* Women who suffer from other functional diseases not related to Musculoskeletal pain.

Ages: 18 Years to 57 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study involved only female gender (N=66) women
Enrollment: 66 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Change in musculoskeletal pain level in the lower back, neck, upper extremities, and lower extremities. | Baseline and Week 12
  Pain levels will be self-reported using the Numeric Rating Scale (NRS-11), a validated 11-point scale ranging from 0 (no pain) to 10 (worst possible pain). Participants will report pain in four body regions: lower back, neck, upper extremities, and lower extremities. The method of assessment was Numeric Rating Scale (NRS-11), administered in-person and via teleconsultation.

SECONDARY OUTCOMES:
Change in flexibility. | Baseline and Week 12
  Flexibility of major joints and muscle groups (especially lower extremities) will be assessed using standard range-of-motion and stretch tests. The method of assessment was manual flexibility tests (sit-and-reach, joint range assessments)
Change in muscle strength in upper and lower extremities and trunk. | Baseline and Week 12
  Muscle strength will be measured using a handheld dynamometer (MicroFET2). Assessments will include trunk flexors/extensors, thigh flexors/extensors, and upper limb muscles (shoulder, elbow, wrist).The method of assessment was Handheld Dynamometer (MicroFET2).

OTHER OUTCOMES:
Change in Body Weight | Baseline and Week 12
  Body weight will be measured using a calibrated digital scale to assess changes over the course of the 12-week intervention. The method of assessment was standard anthropometric measurement tools. The unit of measure: Kilograms per square meter (kg/m²)
Change in body mass index (BMI). | Baseline and Week 12
  BMI will be calculated using measured weight and height, according to the formula: weight (kg) / [height (m)]². This will assess changes in body composition over the course of the 12-week intervention. The method of assessment: was standard anthropometric measurement tools.

CONTACTS AND LOCATIONS:
Overall Officials: Munib Fathe, Principal Investigator — University of Mosul
Locations (1):
- College of Physical Education and Sport Sciences, Mosul, Nineveh Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Data availability will be available on request by contact with corresponding author on email : m.a.fathi@uomsul.edu.iq
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available beginning 6 months after publication and for up to 3 years. Requests will be reviewed by the study's data-sharing committee to ensure alignment with ethical standards and scientific merit.
Access Criteria: Individual Participant Data (IPD) and related supporting documentation (such as the study protocol, statistical analysis plan, and informed consent form) will be made available to qualified researchers upon reasonable request. Access will be granted to researchers affiliated with academic institutions, non-profit organizations, or other recognized research bodies for the purpose of secondary analysis, meta-analysis, or other ethically approved scientific research.
  Requests for access should include a clear research proposal, objectives, and a data use agreement outlining how the data will be protected and used in compliance with applicable ethical and data protection standards.
  To request access, researchers may contact the corresponding author via the email address provided in the publication or through the institutional contact listed in the trial registration. Data will be shared in a de-identified format to ensure participant confidentiality.
URL: https://osf.io/9u2vx/?view_only=daea272a2161482b8dde69fe29d406f0

REFERENCES:
- [Background] Mesa-Castrillon CI, Simic M, Ferreira ML, Bennell KL, Luscombe GM, Gater K, Beckenkamp PR, Michell A, Bauman A, de Luca K, Bunker S, Clavisi O, Ferreira PH. Effectiveness of an eHealth-Delivered Program to Empower People With Musculoskeletal Pain in Rural Australia: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2024 Apr;76(4):570-581. doi: 10.1002/acr.25272. Epub 2024 Jan 29. PMID 37984995
- [Background] Mesa-Castrillon CI, Simic M, Ferreira ML, Hatswell K, Luscombe G, de Gregorio AM, Davis PR, Bauman A, Bunker S, Clavisi O, Knox G, Bennell KL, Ferreira PH. EHealth to empower patients with musculoskeletal pain in rural Australia (EMPoweR) a randomised clinical trial: study protocol. BMC Musculoskelet Disord. 2021 Jan 5;22(1):11. doi: 10.1186/s12891-020-03866-2. PMID 33402161
- [Background] Frattali CM. National Institutes of Health, Warren Grant Magnuson Clinical Center. ASHA. 1999 Jul-Aug;41(4):46-9. No abstract available. PMID 10420662
- [Background] Mesa-Castrillon CI, Beckenkamp PR, Ferreira M, Simic M, Davis PR, Michell A, Pappas E, Luscombe G, Noronha M, Ferreira P. Global prevalence of musculoskeletal pain in rural and urban populations. A systematic review with meta-analysis. Musculoskeletal pain in rural and urban populations. Aust J Rural Health. 2024 Oct;32(5):864-876. doi: 10.1111/ajr.13161. Epub 2024 Jul 4. PMID 38963186
- [Background] Lombard C, Harrison C, Kozica S, Zoungas S, Ranasinha S, Teede H. Preventing Weight Gain in Women in Rural Communities: A Cluster Randomised Controlled Trial. PLoS Med. 2016 Jan 19;13(1):e1001941. doi: 10.1371/journal.pmed.1001941. eCollection 2016 Jan. PMID 26785406
- [Background] Gonzalez-Rocha A, Mendez-Sanchez L, Ortiz-Rodriguez MA, Denova-Gutierrez E. Effect Of Exercise on Muscle Mass, Fat Mass, Bone Mass, Muscular Strength and Physical Performance in Community Dwelling Older Adults: Systematic Review and Meta-Analysis. Aging Dis. 2022 Oct 1;13(5):1421-1435. doi: 10.14336/AD.2022.0215. eCollection 2022 Oct 1. PMID 36186132
- [Background] Allworth I, Luscombe G, Ferreira P, Mesa-Castrillon C. Exploring participant satisfaction with an eHealth intervention for low back pain and knee osteoarthritis: Enhancing physiotherapy access in rural Australia. Musculoskelet Sci Pract. 2025 Apr;76:103252. doi: 10.1016/j.msksp.2024.103252. Epub 2025 Jan 9. PMID 39805211
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Bashshur RL, Shannon GW, Smith BR, Alverson DC, Antoniotti N, Barsan WG, Bashshur N, Brown EM, Coye MJ, Doarn CR, Ferguson S, Grigsby J, Krupinski EA, Kvedar JC, Linkous J, Merrell RC, Nesbitt T, Poropatich R, Rheuban KS, Sanders JH, Watson AR, Weinstein RS, Yellowlees P. The empirical foundations of telemedicine interventions for chronic disease management. Telemed J E Health. 2014 Sep;20(9):769-800. doi: 10.1089/tmj.2014.9981. Epub 2014 Jun 26. PMID 24968105
- [Background] Rockwell KL, Gilroy AS. Incorporating telemedicine as part of COVID-19 outbreak response systems. Am J Manag Care. 2020 Apr;26(4):147-148. doi: 10.37765/ajmc.2020.42784. PMID 32270980
- [Background] Akbar KA, Try P, Viwattanakulvanid P, Kallawicha K. Work-Related Musculoskeletal Disorders Among Farmers in the Southeast Asia Region: A Systematic Review. Saf Health Work. 2023 Sep;14(3):243-249. doi: 10.1016/j.shaw.2023.05.001. Epub 2023 May 13. PMID 37818214
- [Background] Alonso Monteiro Bezerra M, Hellwig N, da Rocha Castelar Pinheiro G, Souza Lopes C. Prevalence of chronic musculoskeletal conditions and associated factors in Brazilian adults - National Health Survey. BMC Public Health. 2018 Feb 27;18(1):287. doi: 10.1186/s12889-018-5192-4. PMID 29482524
- [Background] Walker-Bone K, Palmer KT. Musculoskeletal disorders in farmers and farm workers. Occup Med (Lond). 2002 Dec;52(8):441-50. doi: 10.1093/occmed/52.8.441. PMID 12488514
- [Background] Osborne A, Blake C, McNamara J, Meredith D, Phelan J, Cunningham C. Musculoskeletal disorders among Irish farmers. Occup Med (Lond). 2010 Dec;60(8):598-603. doi: 10.1093/occmed/kqq146. Epub 2010 Sep 15. PMID 20844056
- [Background] Hulshof CTJ, Pega F, Neupane S, Colosio C, Daams JG, Kc P, Kuijer PPFM, Mandic-Rajcevic S, Masci F, van der Molen HF, Nygard CH, Oakman J, Proper KI, Frings-Dresen MHW. The effect of occupational exposure to ergonomic risk factors on osteoarthritis of hip or knee and selected other musculoskeletal diseases: A systematic review and meta-analysis from the WHO/ILO Joint Estimates of the Work-related Burden of Disease and Injury. Environ Int. 2021 May;150:106349. doi: 10.1016/j.envint.2020.106349. Epub 2021 Feb 3. PMID 33546919
- [Background] Ganesh S, Chhabra D, Kumari N. The effectiveness of rehabilitation on pain-free farming in agriculture workers with low back pain in India. Work. 2016 Oct 17;55(2):399-411. doi: 10.3233/WOR-162403. PMID 27689586
- [Background] Fathe MA, Hasan MS, Karash SJ. The Effectiveness of a Rehabilitative Program on the Cervical and Lumbar Pain Relief for Rural Women. Annals of Applied Sport Science. 1 martie 2022;10(1):1-8. https://doi.org/10.52547/aassjournal.985
- Available data/document: Individual Participant Data Set: m.a.fathi@uomosul.edu.iq — https://osf.io/9u2vx/?view_only=daea272a2161482b8dde69fe29d406f0 — De-identified individual participant data is available through the provided OSF link

DOCUMENTS (3):
  • Study Protocol: Decision (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT07129356/Prot_000.pdf
  • Study Protocol: Decision E.A.C (2024-06-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT07129356/Prot_001.pdf
  • Informed Consent Form: L.E.A (2024-06-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT07129356/ICF_002.pdf